CLINICAL TRIAL: NCT07223125
Title: A Phase 1 Study of JNJ-89862175, an Ectonucleotide Pyrophosphatase/Phosphodiesterase Family Member 3 Antibody Drug Conjugate, for Advanced Solid Tumors
Brief Title: A Study of JNJ-89862175 for Treatment of Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 89862175LUC1001; 89862175LUC1001 (Other: Janssen Research & Development, LLC); 2025-521407-52-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-10-30; First posted 2025-10-31 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Advanced-stage Solid Tumors

STUDY DESIGN:
Intervention Model Description: Participants may be randomized in Part 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JNJ-89862175 (Experimental): Participants will receive JNJ-89862175 in Part 1 to determine the recommended phase 2 doses (RP2Ds). Dose-escalation and de-escalation will be based on study evaluation team (SET) decision. In Part 2, participants will receive JNJ-89862175 at the RP2Ds determined in Part 1.
  Interventions: Drug: JNJ-89862175

INTERVENTIONS:
Drug: JNJ-89862175 — JNJ-89862175 will be administered.

SUMMARY:
The purpose of this study is to determine safe and effective dose (recommended phase 2 doses [RP2Ds]) of JNJ-89862175 in Part 1 (dose escalation), and to further evaluate how safe JNJ-89862175 is at the RP2Ds in Part 2 (dose expansion) in participants with advanced stage solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed, metastatic or unresectable solid tumor of lung adenocarcinoma, renal cell carcinoma (RCC): clear cell or papillary carcinoma, endometrioid ovarian cancer and endometrioid uterine carcinoma
* Have an eastern cooperative oncology group (ECOG) performance status of 0 to 1 at screening
* Participants on study drug and for 4 months after the last dose of study drug must not breastfeed or be pregnant, not donate gametes (that is, eggs or sperms) or freeze for future use for the purposes of assisted reproduction and wear an external condom

Exclusion Criteria:

* Active central nervous system (CNS) involvement unless clinically stable
* History of clinically significant cardiovascular disease within 6 months prior to signing informed consent
* History of solid organ or hematologic stem cell transplantation
* Known allergies, hypersensitivity, or intolerance to excipients of JNJ-89862175
* Has prior or concurrent second malignancy (other than the disease under study) in which the natural history or treatment is likely to interfere with safety endpoints or efficacy of the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2028-08-15 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Dose-Limiting Toxicity (DLTs) | Up to 21 days
  The DLTs are specific adverse events that includes high grade hematologic or non-hematologic toxicities with exceptions and/or toxicities leading to treatment discontinuation.
Part 1: Number of Participants with Adverse Events (AEs) by Severity | Up to 2 years and 10 months
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product and does not necessarily have a causal relationship with the intervention. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Part 2: Number of Participants with Adverse Events (AEs) by Severity at RP2D | Up to 2 years and 10 months
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product and does not necessarily have a causal relationship with the intervention. Severity will be graded according to the NCI-CTCAE version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years and 10 months
  ORR is defined as the percentage of participants who have best overall response of complete response (CR) or partial response (PR) according to response evaluation criteria in solid tumors (RECIST) version (v.) 1.1.
Progression Free Survival (PFS) | Up to 2 years and 10 months
  PFS is defined as the time from the first dose of JNJ-89862175 to either disease progression according to RECIST v. 1.1, or death due to any cause, whichever comes first.
Duration of Response (DOR) | Up to 2 years and 10 months
  DOR is defined as the time from the date of initial documentation of a response to the date of first documented evidence of disease progression according to RECIST v. 1.1, or death due to any cause, whichever occurs first.
Maximum Plasma Concentration (Cmax) for JNJ-89862175 (Total and Conjugated Antibody, Free Payload and Major Metabolite) | Up to 2 years and 10 months
  Serum samples will be analyzed to determine Cmax of JNJ-89862175 with total and conjugated antibody, free payload and major metabolite.
Observed Plasma Concentration Immediately Before Next Dose Administration (Ctrough) of JNJ-89862175 (Total and Conjugated Antibody, Free Payload and Major Metabolite) | Up to 2 years and 10 months
  Ctrough of JNJ-89862175 with total and conjugated antibody, free payload and major metabolite will be reported.
Time to Reach Cmax (Tmax) for JNJ-89862175 (Total and Conjugated Antibody, Free Payload and Major Metabolite) | Up to 2 years and 10 months
  Tmax defined as the the time to reach maximum observed plasma concentration of JNJ-89862175 with total and conjugated antibody, free payload and major metabolite will be reported.
Area Under the Plasma Concentration - Time (AUC [0-t]) Curve for JNJ-89862175 (Total and Conjugated Antibody, Free Payload and Major Metabolite) | Up to 2 years and 10 months
  AUC (0-t) defined as area under the plasma concentration-time curve during a dosing interval of JNJ-89862175 with total and conjugated antibody, free payload and major metabolite will be reported.
Accumulation Ratio of JNJ-89862175 (Total and Conjugated Antibody, Free Payload and Major Metabolite) | Up to 2 years and 10 months
  Accumulation ratio of JNJ-89862175 with total and conjugated antibody, free payload and major metabolite will be reported.
Number of Participants With Anti JNJ-89862175 Antibodies | Up to 2 years and 10 months
  Serum samples will be analyzed for the detection of anti-JNJ-89862175 antibodies using a validated assay method.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - AdventHealth Orlando, Orlando, Florida
  - NEXT Oncology, Irving, Texas
- Gustave Roussy, Villejuif, France

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency